CLINICAL TRIAL: NCT06150326
Title: Medical Honey for Wound Treatment in Intensive Care. (MICARéa) Randomized, Controlled, Single-center Pilot Study.
Acronym: MICAREA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A01393-42
Record Dates: First submitted 2023-10-18; First posted 2023-11-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Wound Heal; Critical Illness
Keywords: HONEY
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel arms, single-blinded, single-center study
Who Masked: Outcomes Assessor
Masking Description: The primary outcome is the area of the wound, which will be measured by 3 nurses blinded to the study arm, using a layer of the wound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- medical honey (Experimental): the patients randomised to this arm will have honey (Activon® Advancis Medical.)
  Interventions: Device: medical honey Activon® 25g Tube
- standard of care (Active Comparator): the patients randomised to this arm will have standard of care recommanded by HAS (french organisation)
  Interventions: Device: standard of care

INTERVENTIONS:
Device: medical honey Activon® 25g Tube — no blinding procedures will be set up for the adminisration of the treatement
  Other Names: medical honey
  Arms: medical honey
Device: standard of care — no blinding procedures will be set up for the adminisration of the treatement
  Other Names: recommendation of HAS ( french administration)
  Arms: standard of care

SUMMARY:
Wound management is a real public health issue in France. To date, a wide range of devices exists to treat these wounds, depending on their nature and stage of evolution. Honey has been proposed for the care of wounds and is effective in reducing the surface of wounds and the pain perceived by patients. Inanition, its use is very simple compared to usual care, requiring different types of dressing accross time. In the intensive care unit, patients are prone to suffering or developing numerous types of wound, but the interest of honey has not been investigated yet.

We propose a prospective, monocentric, randomized, single-blind, controlled clinical trial to assess the efficacy of managing acute cutaneous wounds with honey (Activon®) compared with standard care, in intensive care patients. The primary endpoint is the percentage of wound surface area reduction measured at 15 days from inclusion.

DETAILED DESCRIPTION:
Wound management is a real public health issue in France. It affects around 2 million people, and represents a cost of almost 1 billion euros for chronic wounds. Patients in the intensive care unit are prone to suffering or developing numerous types of wound: ulcers, surgical or traumatic wounds on admission or during the stay, pressure sores and wounds associated with medical devices...

Several studies have evaluated the use of honey in chronic and acute wounds. It is effective in reducing wound surface area and decreasing pain perceived by patients. A few randomized controlled studies also show faster wound healing, with a significantly greater reduction in surface area, but these mainly concern chronic wounds with long treatment times. Although medical honey is CE-marked for the treatment of acute wounds, no studies have been carried out on the intensive care patient population. The aim of this study is to assess the efficacy of honey (Activon® , Advancis Medical laboratory - DEODAMED, Saint Die des Vosges - France) in the treatment of wounds occurring in intensive care patients, compared with the use of standard devices.

Critically ill patients with one or more acute wound (ie <8 days), will be included in absence of known allergy to honey and after consent (by the patient of his/her next of kin if he/she is not able to consent). The wound will be randomized to be treated with honey or standerd care, a maximum of 3 wounds will be randomized by patients. A drawing of the wound will be taken using a layer at inclusion, D7 and D15 (or hospital discharge if it happens first). The area of the wound will be measures by 3 nurses, blinded to the treatment arm, using the formula (A=LengthxWidthxπ/4). The patients will be follow-up at 3 months with a on-site visit to record the date of definitive wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in surgical intensive care unit A -USC PTO CHU ANGERS
* Informed consent signed by patient or relative (or emergency inclusion procedure)
* Patient with one or more wounds ≥ 4 cm2, evolving for less than 8 days, including: stage 2, 3, 4 pressure sores, lacerations, ulcers, dermabrasions and scar disunions.

Exclusion Criteria:

* Patients with honey intolerance/allergy to bee stings
* Patients with wounds lasting more than 8 days
* Patient with a bleeding wound,
* Patient with a tunneled wound
* Patients with chronic dermatoses
* Patient with an estimated life expectancy < 15 days
* Expected discharge ≤48 hours.
* No affiliation to a French social security scheme or beneficiary of such a scheme.
* Pregnant, breast-feeding or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
percentage of wound area reduction measured 15 days after inclusion (or on hospital discharge if before Day15). | 15 days
  R = (AJ15-AJ0)/SJ0 x100 with wound area obtained as the mean of the measures made by 3 nurses using a layer of the wound and the formula Area = maximal Length x maximal Width x π/4 R, percentage reduction in surface area (expressed in %); S, surface area (cm²); D, day; D0=day of inclusion

SECONDARY OUTCOMES:
percentage of patient with pain | Day0, Day7 and Day15
  pain evaluation before and after wound care at Day0,Day7 and Day15, using a numerical scale (graduated from 0 to 10) or the Behavior Pain Scale. A scale >3 or a BPS>6 are indicative of significant pain
total healing, | Day0, Day7 and Day15
  to assess total healing, measured by the proportion of patients with total skin healing at Day7, Day15 (or hospital discharge if before Day15) and Day90 (outpatient visit).
scarring progress | Day0, Day7, Day15 and Day90:
  To assess scarring progress at Day0, Day7, Day15 and Day90 using a visual colorimetric scale (black = necrosis; yellow = fibrin; red = budding)
Dressing time | Day0, Day7 and Day15
  To assess the time needed for dressing repair at Day0, Day7 and Day15 (or on day of discharge if before Day15): in minutes
numbers of honey tubes used for dressings | Day0, Day7 and Day15
  to assess Number of honey tubes used for dressings at Day0, Day7 and Day15 (or on day of discharge if before D15).
total honey tubes | Day90
  to asses Number of honey tubes used/returned at Day90 during follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond LASOCKI, MD, PhD, Study Chair — anethesia and critical care department, CHU Angers; catherine ROD, Principal Investigator — anethesia and critical care department, CHU Angers
Locations (1):
- Angers University Hospital, surgical reanimation, Angers, France